CLINICAL TRIAL: NCT03839095
Title: Localized Osteosarcoma of Extremities: Developing a Clinical Prediction Model From a Country With Limited Resources
Brief Title: Localized Osteosarcoma in Upper Egypt: A Clinical Prediction Model
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer, Pediatric Oncology Department, Assiut University
Other Study IDs: IRB_Os_Pred_Mod
Record Dates: First submitted 2019-02-09; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Bone Neoplasms
Keywords: Nonmetastatic Osteosarcoma; Pediatric Cancer; Limb Salvage; Prediction Model
MeSH Terms: conditions — Bone Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
To assess survival outcome of pediatric patients with localized osteosarcoma of the extremities in Upper Egypt, identify factors of prognostic significance for survival, and to determine factors predictive of surgical methods employed in these patients, and developing a clinical model for risk prediction.

DETAILED DESCRIPTION:
Background Osteosarcoma is the most common of all primary malignant bone tumors. Accounting for about 2.6% of all pediatric neoplasms, it predominantly occurs in the extremities, with a peak incidence in the second decade of life.

In Upper Egypt, we have a higher proportion of the population in underdeveloped communities with limited access to medical care so the patients usually seek medical advice at advanced stage leading to a higher prevalence of metastatic disease at initial presentation, as well as a greater proportion of larger tumor size that more likely to be associated with potential adverse risk criteria prior to surgery.

A previous study from Upper Egypt showed that a metastatic disease at diagnosis was independently correlated to a dismal outcome. Since the effect of many other factors of prognostic significance, such as, gender, age, tumor location and response to chemotherapy may have been mitigated by the large effect of the metastatic disease on the prognosis; So, here, we will analyze the data of 30 patients with non-metastatic osteosarcoma of the extremities, to determine prognostic factors associated with survival, and also to develop a model for a better prediction of factors correlated to that a certain surgical approach was employed in these patients based on their baseline clinical data and the tumor response to chemotherapy.

Patients & Methods We will carry out a retrospective analysis of data assembled from medical records of 30 pediatric patients with a histologically-verified non-metastatic osteosarcoma of the extremities treated at South Egypt Cancer Institute with a unified chemotherapy protocol between January 2001 and December 2015. These data will be categorized according to demographic data, clinical characteristics, tumor response to chemotherapy, and surgical methods employed in these patients. Prognostic factors will be determined using univariable and multivariable methods. A predictive model for surgical outcomes in these patients based on the baseline clinical factors, and their tumor response to chemotherapy will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than 19 years.
* Patients diagnosed with verified osteosarcoma involving the extremities.

Exclusion Criteria:

* Patients whose age more than 19 years.
* Non-extremities Osteosarcoma .

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 30 pediatric patients with a histologically-verified non-metastatic osteosarcoma of the extremities treated at South Egypt Cancer Institute with a unified chemotherapy protocol between January 2001 and December 2015.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-08-25 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of treatment initiation until the date of death from any cause or patients censored at last follow up, whichever came first, assessed up to 60 months
  Participants will be retrospectively followed forward in time from the date of initiation of treatment till death from any cause, an expected average of 5 years
Metastasis-Free survival (MFS) | From date of treatment initiation until the date of first documented systemic recurrence or patients censored at last follow up, whichever came first, assessed up to 60 months
  Participants will be retrospectively followed forward in time from the date of initiation of treatment till the occurrence of systemic recurrence, an expected average of 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Morsy AM, Abdelgawad MI, Ahmed BM, Rezk KM, Aboelgheit AM, Ramadan IK, Kamel HEM, Fouad DM, Herdan RA, Shabaan SH, Eltyb HA. Pediatric Osteosarcoma of Extremities: A 15-year Experience From a Tertiary Care Cancer Center in Upper Egypt. J Pediatr Hematol Oncol. 2019 Aug;41(6):e371-e383. doi: 10.1097/MPH.0000000000001407. PMID 30629005